CLINICAL TRIAL: NCT03925506
Title: Identification of Predictive Factors of Inadequate Bowel Preparation in Inpatients. The Quality-In-Patients Study (QIPS)
Brief Title: Predictive Factors of Inadequate Bowel Preparation in Inpatients
Acronym: QIPS
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Lorenzo Fuccio, Professor of Gastroenterology, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: QIPS observational study
Record Dates: First submitted 2019-04-16; First posted 2019-04-24 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Bowel Preparation Solutions; Colonoscopy; Inpatient

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
About 50-70% only of inpatients who undergo colonoscopy have an adequate bowel cleansing, which is far below the recommended threshold of 90%. Variables associated to inadequate colon preparation have not been assessed yet. Identifying such variables would allow to augment the diagnostic yield of colonoscopy, and also to reduce costs related to the need to repeat colonoscopy. Aim of the present study is to find variables independently associated to an inadequate bowel cleansing and to subsequently build and validate a predictive model, which could prove useful in clinical practice to identify hard-to-prepare inpatients. Secondary endpoints are (i) to assess the proportion of patients with inadequate colon cleansing, (ii) to run a cost-effectiveness analysis between patients with adequate cleansing and patients who need to repeat colonoscopy. Patients undergoing urgent colonoscopy, and patients who take the preparation at home will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient ≥18 y.o. who are scheduled elective colonoscopy during hospitalization irrespective of the indication.

Exclusion Criteria:

* Urgent colonoscopy
* Patients who are not hospitalized when taking bowel preparation or when undergoing colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in 12 Centers in Italy, who are scheduled elective colonoscopy irrespective of the indication.
Sampling Method: Non-Probability Sample
Enrollment: 1658 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Inadequate bowel cleansing rate | At the end of the study, 3 months after the beginning of the study.
  The number of inpatients with inadequate bowel preparation over the total number of patients enrolled. Bowel prep will be assessed according to the Boston Bowel Preparation Scale (BBPS). A score less than 2 at one segment of the colon will be considered as inadequate bowel preparation.

SECONDARY OUTCOMES:
Rate of patients scheduled for colonoscopy repetition due to inadequate bowel preparation | At the end of the study, 3 months after the beginning of the study.
  Total number of patients scheduled for repeating colonoscopy over the total number of patients enrolled scheduled for repeating colonoscopy due to poor bowel pre.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Sant'Orsola-Malpighi, Bologna, Italy

REFERENCES:
- [Derived] Fuccio L, Frazzoni L, Spada C, Mussetto A, Fabbri C, Manno M, Aragona G, Zagari RM, Rondonotti E, Manes G, Occhipinti P, Cadoni S, Bazzoli F, Hassan C, Radaelli F; QIPS study group. Factors That Affect Adequacy of Colon Cleansing for Colonoscopy in Hospitalized Patients. Clin Gastroenterol Hepatol. 2021 Feb;19(2):339-348.e7. doi: 10.1016/j.cgh.2020.02.055. Epub 2020 Mar 18. PMID 32200083